CLINICAL TRIAL: NCT01146860
Title: A Multi-centre, Double-blind, Placebo-controlled, Randomised, Parallel Group Study to Assess the Efficacy and Safety of a Herbal Medicinal Product (Dry Extract BNO 1016) in Patients With Acute Rhinosinusitis
Brief Title: Efficacy and Safety of a Herbal Medicinal Product (Dry Extract BNO 1016) in Patients With Acute Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARhiSi-2; 2009-016682-28 (EudraCT Number)
Record Dates: First submitted 2010-06-07; First posted 2010-06-22 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: Acute Rhinosinusitis
Keywords: BNO 1016, acute rhinosinusitis
MeSH Terms: interventions — BNO 1016; Sinupret

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BNO 1016 (Experimental): sugar coated tablets with dry extract (80 mg) of 5 herbal drugs; dosage: 480 mg per day (2 tablets t.i.d.) duration: 15 days
  Interventions: Drug: BNO 1016
- Placebo (Placebo Comparator): sugar coated tablets with identical appearance to active treatment; frequency: 2 tablets t.i.d. duration: 15 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BNO 1016 — sugar coated tablets with dry extract (80 mg) of 5 herbal drugs; dosage: 480 mg per day (2 tablets t.i.d.) duration: 15 days
  Other Names: Sinupret extract
  Arms: BNO 1016
Drug: Placebo — sugar coated tablets with identical appearance to active treatment; frequency: 2 tablets t.i.d. duration 15 days
  Other Names: Placebo to BNO 1016
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the dry extract BNO 1016 is effective and safe in the treatment of acute rhinosinusitis in adults.

DETAILED DESCRIPTION:
The aim of this clinical study is to investigate the efficacy of a 15-days treatment with the herbal medicinal product BNO 1016 for therapy of acute rhinosinusitis in adult patients. Due to the considerable morbidity and the diminished quality of life experienced by people afflicted with acute rhinosinusitis an important aim of the treatment is to reduce the severity of rhinosinusitis symptoms and the duration of the disease. By grading the severity of the disease on the basis of the 5 main rhinosinusitis symptoms the investigator will assess the efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of acute rhinosinusitis

* characterized by a major symptom score (MSS) ≥ 8 and ≤ 12 points (minimum 0, maximum 15 points)
* individual score for facial pain/pressure ≥ 1 (mild) and ≤ 2 (moderate)
* confirmed by ultrasonography of paranasal sinuses
* with presence of symptoms ≤ 3 days prior to inclusion

Exclusion Criteria:

* Chronic rhinosinusitis
* Polyposis nasi
* Anatomical deviations of the nasal septum that significantly impair nasal and paranasal ventilation/airflow
* Acute symptoms of a known allergic rhinitis
* Patients with asthma who have a history of exacerbations within 30 days prior to study inclusion
* Signs or symptoms of fulminant bacterial sinusitis
* Odontogenic sinusitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Jund, MD, Study Chair — Specialist in Otorhinolaryngology
Locations (1):
- Dr. Rainer Jund, Specialist in Otorhinolaryngology, Puchheim, Germany

REFERENCES:
- [Derived] Jund R, Mondigler M, Steindl H, Stammer H, Stierna P, Bachert C; ARhiSi II study group. Clinical efficacy of a dry extract of five herbal drugs in acute viral rhinosinusitis. Rhinology. 2012 Dec;50(4):417-26. doi: 10.4193/Rhino.12.015. PMID 23193534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2010 to April 2010 37 centres (16 ENT and 21 specialists in internal medicine and general practitioners
Groups:
- BNO 1016: sugar coated tablets with dry extract (80 mg) of 5 herbal drugs; daily dose: 480 mg (2 tablets tid)
- Placebo: sugar coated tablets of identical appearance to active treatment
Period: Overall Study
Arm/Group | BNO 1016 | Placebo
Started | 194 | 192
Completed | 194 | 191
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- BNO 1016; Placebo: sugar coated tablets
- Total: Total of all reporting groups
Arm/Group | BNO 1016 | Placebo | Total
Number analyzed (Participants) | 194 | 192 | 386
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 174 | 182 | 356
  >=65 years | 20 | 10 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 41.0 (15.4) | 40.4 (14.3) | 40.7 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 122 | 249
  Male | 67 | 70 | 137
Region of Enrollment [Number; unit: participants]
  Germany | 194 | 192 | 386

OUTCOME MEASURES:

1. Primary Outcome: Major Symptom Score (MSS) Assessed by the Investigator
Description: MSS: sum of the 5 main rhinosinusitis symptoms which are: rhinorrhea (anterior discharge), postnasal drip, nasal congestion, headache, facial pain/pressure.
  Each symptom is individually evaluated using the following 4-point rating scale (scoring system): 0 = none/not present, 1 = mild, 2 = moderate, 3 = severe.
  Thus the MSS ranges from a minimum of 0 to a maximum of 15 score points.
Time Frame: 14 days
Population: FAS: randomised patients with at least one documented application of the drug and post-baseline efficacy data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BNO 1016 | Placebo
Number analyzed (Participants) | 190 | 190
units on a scale | 2.38 (0.18) | 3.41 (0.24)

2. Secondary Outcome: SNOT 20 Symptom Scores
Description: Sino-Nasal Outcome Test (SNOT 20): 20 item questionnaire to assess the symptoms and emotional and social consequences of rhinosinusitis. The symptoms are assessed by the patient using a 6-point rating scale: 0 = not present / no problem, 1 = very mild problem, 2 = mild or slight problem, 3 = moderate problem, 4 = severe problem, 5 = problem as "bad as it can be".
  range: 0 to 100
Time Frame: 14 days
Population: FAS: randomised patients with at least one documented application of the drug and post-baseline efficacy data
Measure: Mean (Standard Deviation); unit: units on a scale (range: 0 - 100)
Arm/Group | BNO 1016 | Placebo
Number analyzed (Participants) | 190 | 190
units on a scale (range: 0 - 100) | 11.02 (12.72) | 15.76 (16.26)

3. Secondary Outcome: Major Symptom Score Assessed by the Patient
Description: as for outcome 1
Time Frame: 14 days
Population: FAS: randomised patients with at least one documented application of the drug and post-baseline efficacy data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BNO 1016 | Placebo
Number analyzed (Participants) | 190 | 190
units on a scale | 2.62 (0.21) | 3.48 (0.24)

4. Secondary Outcome: Percentage of Patients Classified as Responders by the Investigator on a 4-point Rating Scale
Description: General assessment of efficacy using a 4-point rating scale (symptoms healed, improved, unchanged, deteriorated). Patients whose symptoms are improved or healed will be classified as "responders" to treatment. Patients whose symptoms are unchanged or deteriorated as classified as "non-responders".
Time Frame: 14 days
Population: FAS: randomised patients with at least one documented application of the drug and post-baseline efficacy data
Measure: Number; unit: percentage of patients
Arm/Group | BNO 1016 | Placebo
Number analyzed (Participants) | 190 | 190
percentage of patients | 94.2 | 87.4

5. Secondary Outcome: Ultrasonography of Paranasal Sinuses
Description: Percentage of patients with signs of acute rhinosinusitis in ultrasonography of paranasal sinuses will be evaluated. Ultrasonography scans will be visually evaluated by the investigator for signs of rhinosinusitis.
Time Frame: 14 days
Population: FAS: randomised patients with at least one documented application of the drug and post-baseline efficacy data
Measure: Number; unit: percentage of patients
Arm/Group | BNO 1016 | Placebo
Number analyzed (Participants) | 190 | 190
percentage of patients | 26.8 | 38.4

ADVERSE EVENTS:
Arm/Group | BNO 1016 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/194 | 0/191
Other Adverse Events (participants affected / at risk) | 19/194 | 27/191
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNO 1016 (N=194) | Placebo (N=191)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal upper pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3)
Facial pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
ASAT increased (Investigations) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Genital discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Headache and facial pain are rated by investigator based on the description of the patient. This was done to ensure a uniform rating of symptom severity across the investigational sites but nevertheless subjective and open to error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No